CLINICAL TRIAL: NCT02827435
Title: Acute Pharmacokinetic-pharmacodynamic Change of Rocuronium After Reperfusion of Renal Graft During Kidney Transplantation
Brief Title: Acute Pharmacokinetic-pharmacodynamic Change of Rocuronium After Reperfusion of Renal Graft
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chul-Woo Jung, Associate professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Roc_KTPL_PKPD
Record Dates: First submitted 2016-06-14; First posted 2016-07-11 (Estimated); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: End Stage Renal Disease; Transplantation
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Rocuronium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rocuronium bolus (Experimental): rocuronium bromide 1st bolus 0.1mg/kg, rocuronium bromide 2nd bolus 0.4mg/kg
  Interventions: Drug: Rocuronium bromide

INTERVENTIONS:
Drug: Rocuronium bromide — Pharmacokinetic-pharmacodynamic modeling blood sampling and Rocuronium bromide concentration measure muscle relaxation evaluation

SUMMARY:
Reperfusion of renal graft in kidney transplantation can change the pharmacokinetic-pharmacodynamic (PKPD) parameters of rocuronium. The immediate increase of urine output during surgery may change the PKPD parameters of the drugs, including elimination rate. The goal of this study is to characterize the PKPD model of rocuronium during kidney transplantation and establish a basis for adequate dosage of rocuronium in kidney transplantation.

Through PKPD modeling, the changes during reperfusion of the renal graft will be evaluated. Furthermore, the factors related to the changes will be assessed. Adjusting the infusion rate according to the step of kidney transplantation will lead to stable muscle relaxation and fast recovery.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for elective living donor kidney transplantation
* end stage renal disease with oliguria or anuria
* normal BMI (BMI 18.5 ~ 25)
* obtained informed consent

Exclusion Criteria:

* patient with underlying neuromuscular disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2016-07-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
rocuronium plasma concentration (mcg/ml) | 0, 1, 3, 5, 10, 30, 60, 90, 120 minutes after rocuronium second bolus injection
  PKPD modeling from measuring plasma rocuronium concentration and excreted urine rocuronium amount
acceleromyography data (TOF ratio %) | intraoperative
  Muscle relaxation level (TOF, T1) will be evaluated via acceleromyography. The pharmacodynamic modeling with NONMEM throughout the kidney transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Chul-Woo Jung, MD. PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No